CLINICAL TRIAL: NCT02541721
Title: An Open-label Study to Investigate the Effectiveness in Clinical Symptomatic Control and Tolerability of Medical Device LabiaStick#01 in Subjects With Symptomatic Non-hypertrophic Chronic Vulvar Dermatoses
Brief Title: Effectiveness and Tolerability of LabiaStick#01 in Subjects With Symptomatic Non-hypertrophic Chronic Vulvar Dermatoses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New study design will be made
Sponsor: Health Products Research and Development Lda. (Other)
Collaborators: Blueclinical, Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LF-01-01
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Chronic Disease of Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LabiaStick#01 (Experimental): Each participant will have an at least 2-week baseline period followed by a 4-week treatment period with LabiaStick#01.
  Interventions: Device: LabiaStick#01

INTERVENTIONS:
Device: LabiaStick#01 — This medical device has emollient agents whose main function is to increase the skin hydration, provide physical protection and decrease the symptoms and possibility of recurrence of vulvar dermatoses.
  The medical device should be applied once daily, in the evening, after a gentle washing (plain water with no cleansing products), on the affected non-hairy vulvar area.

SUMMARY:
The current study aims to investigate the effectiveness in clinical symptomatic control and tolerability of LabiaStick#01 in women with symptomatic non-hypertrophic chronic vulvar dermatoses.

DETAILED DESCRIPTION:
Vulvar dermatoses are skin disorders that affect the vulva, causing pruritus, irritation and pain. Although the prevalence of these disorders is unknown, it is well accepted that the vulvar symptoms are a common problem for women.

LabiaStick#01 has emollient agents whose main function is to increase the skin hydration, provide physical protection and decrease the symptoms and possibility of recurrence of vulvar dermatoses.

The medical device should be applied once daily, in the evening, after intimal hygiene care.

The primary objective of this study is to evaluate the effectiveness of LabiaStick#01 on the relief of pruritus caused by symptomatic non-hypertrophic chronic vulvar dermatoses.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent.
* Woman, with 18 or more years.
* Diagnosed with symptomatic non-hypertrophic chronic vulvar dermatoses.
* A pruritus score of at least 20 on a 100-mm VAS-PR.
* Willing and able to comply with the study requirements.
* Participant of childbearing potential agrees to remain abstinent or to use an acceptable contraceptive measure for the entire duration of the study.
* Participant not of childbearing potential (e.g., is not sexually active, whose current partner is not of reproductive potential).

Exclusion Criteria:

* Received systemic immunosuppressant therapy (e.g. systemic corticosteroids) within 4 weeks prior to admission.
* Treated with daily topical therapy (e.g. topical corticosteroids, pimecrolimus, and tacrolimus) at the target vulvar area within 2 weeks prior to admission, which in the opinion of the investigator might compromise study results.
* Immunocompromised (e.g., lymphoma, AIDS, Wiskott-Aldrich Syndrome) or have an uncontrolled malignant disease.
* Suffers from systemic or generalized infections (bacterial, viral or fungal).
* Diagnosis of psoriasis, candidiasis, vulvar intraepithelial neoplasia or carcinoma of the vulva.
* Pregnancy or breastfeeding.
* Documented and consistent history of hypersensitivity reactions to similar topical products.
* Any condition that in the opinion of the investigator might prevent the subject from completing the study or interfere with the interpretation of the study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-09; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Reduction on subject's vulvar pruritus score | 14 days during run-in period and 14 days during treatment period
  Reduction on subject's vulvar pruritus score assessed on a 100-mm Visual Analogue Scale for Pruritus Relief (VAS-PR) following once-daily application of LabiaStick#01, for 4 weeks.

SECONDARY OUTCOMES:
Reduction on subject's vulvar burning sensation score | During 4 weeks
  Reduction on subject's vulvar burning sensation score assessed on a 100-mm Visual Analogue Scale (Burning VAS).
Clinical Global Impression of Change (CGI-C) | At Visit 3 (28 days after the end of baseline)
Patient Global Impression of Change (PGI-C) | At Visit 3 (28 days after the end of baseline)
Subjects' opinion on the acceptability of the medical device | At Visit 3 (28 days after the end of baseline)
  Subjects' opinion on the acceptability of the medical device (cosmetic acceptability and easiness of use)
Need of rescue medication | Up to 6 weeks
Adverse events | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: José Martinez de Oliveira, MD, PhD, Principal Investigator — HPRD
Locations (6):
- Portugal (6):
  - Hospital Garcia da Orta, EPE, Lisbon, Almada
  - Centro Hospitalar Cova da Beira EPE, Covilha, Castelo Branco District
  - Apomédica - Serviços Médicos Ltd, Póvoa de Varzim, Porto District
  - Unidade Local de Saúde de Matosinhos, Matosinhos Municipality, Senhora Da Hora
  - Centro Hospitalar de S. João EPE, Porto
  - Centro Hospitalar Vila Nova de Gaia/Espinho, E.P.E, Vila Nova de Gaia